CLINICAL TRIAL: NCT01791855
Title: A PHASE 1, SINGLE DOSE, OPEN-LABEL STUDY TO EVALUATE THE EFFECT OF RENAL IMPAIRMENT ON THE PHARMACOKINETICS OF PF-04634817
Brief Title: PF-04634817 Renal Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B1261008; 2013-000360-29 (EudraCT Number)
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-08

CONDITIONS: Renal Insufficiency
Keywords: Subjects with Renal Impairment; healthy
MeSH Terms: conditions — Renal Insufficiency | interventions — PF-04634817

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy Volunteers (Experimental)
  Interventions: Drug: PF-04634817
- Mild Renal Impairment (Experimental)
  Interventions: Drug: PF-04634817
- Moderate renal impairment (Experimental)
  Interventions: Drug: PF-04634817
- Severe renal impairment (Experimental)
  Interventions: Drug: PF-04634817

INTERVENTIONS:
Drug: PF-04634817 — Single 50 mg dose administered to subjects with normal renal function (creatinine clearance greater than or equal to 90 ml/min)
  Arms: Healthy Volunteers
Drug: PF-04634817 — Single 50 mg dose administered to subjects with mild renal impairment (creatinine clearance 60-89 ml/min)
  Arms: Mild Renal Impairment
Drug: PF-04634817 — Single 50 mg dose administered to subjects with moderate renal impairment (creatinine clearance 30-59 ml/min)
  Arms: Moderate renal impairment
Drug: PF-04634817 — Single 50 mg dose administered to subjects with severe renal impairment (creatinine clearance 15-29 ml/min)
  Arms: Severe renal impairment

SUMMARY:
Patients with renal impairment are the target population for PF-04634817. The clearance mechanism of this drug means that exposure may be increased in subjects with renal impairment. This study will investigate the effect of the drug in subjects with varying degrees of renal impairment. Pharmacokinetics, safety and toleration will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (non child bearing potential aged 18-75 years
* Documented renal impairment (mild, moderate or severe using Cockcroft-Gault equation) or matched healthy volunteers (age, weight and gender)

Exclusion Criteria:

* Subjects with acute renal failure
* Subjects receiving, or likely to receive, CYP450 3A4 inhibitors
* Abnormal ECG at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-05-10 (Actual); Primary Completion 2013-09-03 (Actual); Study Completion 2013-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Avail Clinical Research, LLC, DeLand, Florida
  - Unversity of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Tesch GH, Pullen N, Jesson MI, Schlerman FJ, Nikolic-Paterson DJ. Combined inhibition of CCR2 and ACE provides added protection against progression of diabetic nephropathy in Nos3-deficient mice. Am J Physiol Renal Physiol. 2019 Dec 1;317(6):F1439-F1449. doi: 10.1152/ajprenal.00340.2019. Epub 2019 Sep 30. PMID 31566438
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1261008&StudyName=PF-04634817%20Renal%20Impairment%20Study

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Renal Function: An oral dose of PF-04634817 50 milligram (mg) was administered to participants with normal renal function (defined as a creatinine clearance [CrCL] of more than or equal [>=] to 90 milligrams [mL]/minute [min], estimated using the Cockcroft-Gault Equation).
- Mild Renal Impairment: An oral dose of PF-04634817 50 mg was administered to participants with mild renal impairment (defined as a CrCL of 60 to 89 mL/min, estimated using the Cockcroft-Gault Equation).
- Moderate Renal Impairment: An oral dose of PF-04634817 50 mg was administered to participants with moderate renal impairment (defined as a CrCL of 30 to 59 mL/min, estimated using the Cockcroft-Gault Equation).
- Severe Renal Impairment: An oral dose of PF-04634817 50 mg was administered to participants with severe renal impairment (defined as a CrCL of 15 to 29 mL/min, estimated using the Cockcroft-Gault Equation).
Period: Overall Study
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Started | 8 | 9 | 8 | 7
Treated | 8 | 8 | 8 | 7
Completed | 8 | 8 | 8 | 6
Not Completed | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Randomized, not treated | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis included the participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Total
Number analyzed (Participants) | 8 | 8 | 8 | 7 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (5.2) | 66.5 (3.9) | 61.9 (3.2) | 59.0 (12.0) | 61.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 3 | 12
  Male | 5 | 4 | 6 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to 48 Hours[AUC (0 - 48)]
Description: AUC (0 - 48)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to 48hours.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 16, 24, 32, 40, 48, 56, 64, 72, 84, 96, 108, 120, 132, 144, 156, 216, 312 hours post dose
Population: The pharmacokinetics (PK) parameter analysis population was defined as all participants randomized and treated who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter (ng*h/mL)
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 7
Nanogram*hour/milliliter (ng*h/mL) | 1294 (27) | 1399 (42) | 2024 (35) | 2860 (34)

2. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: as for outcome 1
Population: The PK parameter analysis population was defined as all participants randomized and treated who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 7
ng*h/mL | 1467 (29) | 1575 (44) | 2610 (42) | 3845 (37)

3. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - Inf)]
Description: AUC (0 - inf)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time.
Time Frame: as for outcome 1
Population: The PK parameter analysis population was defined as all participants randomized and treated who had at least 1 of the PK parameters of primary interest. N = number of participants with reportable AUC(0-inf) values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 7 | 7
ng*h/mL | 1473 (29) | 1584 (44) | 2611 (45) | 3877 (37)

4. Primary Outcome: Apparent Oral Clearance (CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: as for outcome 1
Population: The PK parameter analysis population was defined as all participants randomized and treated who had at least 1 of the PK parameters of primary interest. N = the number of participants with reportable CL/F values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/minute (mL/min)
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 7 | 7
milliliter/minute (mL/min) | 565.8 (29) | 526.8 (44) | 319.2 (45) | 215.2 (37)

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 7
ng/mL | 124.6 (49) | 111.4 (66) | 123.7 (59) | 132.3 (59)

6. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 7
hours | 2.01 [1.50 to 3.00] | 2.50 [1.00 to 8.00] | 2.00 [1.50 to 8.00] | 3.00 [1.00 to 12.0]

7. Primary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: as for outcome 1
Population: The PK parameter analysis population was defined as all participants randomized and treated who had at least 1 of the PK parameters of primary interest. N = the number of participants with reportable Vz/F values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 7 | 7
Liter (L) | 1453 (35) | 1808 (38) | 1162 (57) | 742.3 (53)

8. Primary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 1
Population: The PK parameter analysis population was defined as all participants randomized and treated who had at least 1 of the PK parameters of primary interest. N = the number of participants with reportable t1/2 values.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 7 | 7
hours | 31.01 (11.33) | 43.94 (24.40) | 43.57 (11.89) | 44.94 (23.96)

9. Secondary Outcome: Amount of Unchanged Drug Excreted in Urine Over 48 Hours (Ae48)
Description: Amount of unchanged drug excreted in urine over 48 hours (Ae48) = urine concentration x volume of urine.
Time Frame: 0-24, 24-48 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 7
ng | 9303000 (48) | 5993000 (47) | 4997000 (26) | 3097000 (65)

10. Secondary Outcome: Percentage of the Dose Excreted Unchanged in the Urine Over 48 Hours (Ae48%)
Description: Percentage (%) of drug excreted unchanged in urine over 48 hours (Ae48%) = Ae48/(dose x 100).
Time Frame: 0-24, 24-48 post dose
Population: The PK parameter analysis population was defined as all participants randomized and treated who had at least 1 of the PK parameters of primary interest. Note that the measure of dispersion should be simply coefficient of variation (CV) instead of geometric CV (GCV) for Ae48%. GCV was chosen due to absence of CV in the options given for that field.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of unchanged drug excreted
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 7
percentage of unchanged drug excreted | 18.61 (44) | 12.00 (43) | 9.989 (25) | 6.193 (62)

11. Secondary Outcome: Renal Clearance Over a 48-hour Interval(CLr48)
Description: Renal clearance over a 48-hour interval (CLr48) = Ae48/AUC48.
Time Frame: 0-24, 24-48 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 7
mL/min | 119.8 (39) | 71.40 (41) | 41.13 (36) | 18.05 (59)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 1/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Renal Function (N=8) | Mild Renal Impairment (N=8) | Moderate Renal Impairment (N=8) | Severe Renal Impairment (N=7)
Pyrexia (General disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Renal Function (N=8) | Mild Renal Impairment (N=8) | Moderate Renal Impairment (N=8) | Severe Renal Impairment (N=7)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Designation of primary and secondary endpoints was based on the discretion of the study team, as the endpoints were not characterized clearly in the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.